CLINICAL TRIAL: NCT02586142
Title: Botulinum Toxin Injections by Ultrasounds Guidance and Stretching Exercise in Spastic Toe Clawing
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NMRPG890041
Record Dates: First submitted 2015-10-12; First posted 2015-10-26 (Estimated); Last update posted 2015-10-26 (Estimated); Status verified 2010-08

CONDITIONS: Cerebrovascular Accident
Keywords: spasticity; claw toe; ultrasounds guidance; botulinum toxin; stretching exercise
MeSH Terms: conditions — Stroke; Muscle Spasticity; Hammer Toe Syndrome | interventions — Botulinum Toxins, Type A; Botulinum Toxins; Muscle Stretching Exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Botulinum toxin type A(BTX-A) injection (Experimental): To inject Botulinum toxin type A on the spasticity lower extremities for participants by ultrasounds guidance.
  Interventions: Drug: Botulinum Toxin Type A
- BTX-A injection plus stretching exercise (Active Comparator): Inject Botulinum toxin type A on the spasticity lower extremity for participants by ultrasounds guidance. After injection, arrange them to receive stretching exercise in Kaoshiung Chang Gung Memorial Hospital 3 time per week for 3 months.
  Interventions: Drug: Botulinum Toxin Type A; Other: Stretching exercise

INTERVENTIONS:
Drug: Botulinum Toxin Type A — To inject Botulinum toxin type A on the spasticity lower extremity for stroke patients by ultrasounds guidance.
  Other Names: Botulinum toxin
Other: Stretching exercise — After accepting Botulinum toxin type A injection, participants will be arranged to receive stretch exercise in Kaohsiung Chang Gung Memorial Hospital 3 times per week, for 3 month.
  Arms: BTX-A injection plus stretching exercise

SUMMARY:
Claw toes deformity result in spasticity often seem in patients with central nerve disease. It also cause pressure sore in foot and pain during walking that didn't well improve under traditional treatment. There are few relative reports about the Botulinum toxin type A (BTX-A) injection on claw toe. The investigators' study has two main purposes:

1. assess the efficiency of BTX-A injection under ultrasonographyic guidance on improving lower extremities function, pain and spasticity in patients with symptomatic claw toes.
2. assess if regular stretching exercise can strength the efficiency of BTX-A injection on improving lower extremities function, pain and spasticity.

DETAILED DESCRIPTION:
The investigators will enroll 50 hemiplegic stroke patients met the inclusion criteria(onset more than 6 month, lower extremity Brunnstrome stage more than stage IV, walking without assistance devices and pain during walking due to claw toe. The investigators will focus and inject BTX-A with ultrasonographyic guidance on flexor digitorum longus and brevis(both 50 unit). If patients combine ankle plantar flexors spasticity, the investigators will inject another 50 unit on both the medial and lateral head of gastrocnemius . Every patients will receive regular stretching exercise in hospital and do self stretching exercise at home for 3 months after injection. Patients will be evaluated at 2 weeks, 4 weeks and 12 weeks, 24 weeks and 1 year after injection. Outcome measure include severity of spasticity and pain, sensory and motor function, range of motion, functional assessment of lower extremity and analyze pressure under foot.

ELIGIBILITY:
Inclusion Criteria:

* Patient with spasticity toe clawing(metatarsophalange jointextension, proximal and distal phalange joint flexion)
* MAS scale of metatarsophalange joint and interphalangeal joint more than 2
* Pain during walking, abnormal gait patterns and can't wear shoess due to claw toe
* Haven't received botox or phenol or alcohol injections before

Exclusion Criteria:

* Lower extremities joint contrature, bone deformity
* Had received botox injections or phenol injections or before due to lower extremities spasticity
* Combine other neuromuscular system disease
* Severe cognition disorder or aphasia after stroke
* Significant atrophy of flexor digitorum longus and brevis
* Allergy to botox
* Infection on injection site
* Have systemic infection
* Now accept aminioglycoside or other medicine will affect neuromusclar transition

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-08; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Spasticity severity scale | Change from Baseline data at 1 year
  patients will be evaluated at 4 weeks, 8 weeks, 12 weeks, 24 weeks and 1 year after injection 0=none, 1=mild, 2= median, 3=severe

SECONDARY OUTCOMES:
Sensory function scale | Change from Baseline data at 1 year
  patients will be evaluated at 4 weeks, 8 weeks, 12 weeks, 24 weeks and 1 year after injection 0=no feeling, 1=abnormal, 2= normal
Brunnstrome stage | Change from Baseline data at 1 year
  patients will be evaluated at 4 weeks, 8 weeks, 12 weeks, 24 weeks and 1 year after injection
Manual muscle test | Change from Baseline data at 1 year
  patients will be evaluated at 4 weeks, 8 weeks, 12 weeks, 24 weeks and 1 year after injection including toe flexion/ extension, ankle plantar flexion/ dorsiflexion
Functional ambulation classification scale | Change from Baseline data at 1 year
  patients will be evaluated at 4 weeks, 8 weeks, 12 weeks, 24 weeks and 1 year after injection
Active range of motion measured by goniometer | Change from Baseline data at 1 year
  patients will be evaluated at 4 weeks, 8 weeks, 12 weeks, 24 weeks and 1 year after injection
Modified Ashworth scale(MAS) | Change from Baseline data at 1 year
  patients will be evaluated at 4 weeks, 8 weeks, 12 weeks, 24 weeks and 1 year after injection
Pain severity measurement recorded by VAS | Change from Baseline data at 1 year
  patients will be evaluated at 4 weeks, 8 weeks, 12 weeks, 24 weeks and 1 year after injection 0=no pain; 100=maximum
To develop a questionnaire (ABILOCO questionnaire) | Change from Baseline data at 1 year
  patients will be evaluated at 4 weeks, 8 weeks, 12 weeks, 24 weeks and 1 year after injection.
  Its a Rasch-built 13-item questionnaire to assess locomotion ability in stroke patients.
Berg Balance test | Change from Baseline data at 1 year
  patients will be evaluated at 4 weeks, 8 weeks, 12 weeks, 24 weeks and 1 year after injection
Get up and go test | Change from Baseline data at 1 year
  patients will be evaluated at 4 weeks, 8 weeks, 12 weeks, 24 weeks and 1 year after injection
10-meter walking test | Change from Baseline data at 1 year
  patients will be evaluated at 4 weeks, 8 weeks, 12 weeks, 24 weeks and 1 year after injection
Fugl-Meyer Assessment | Change from Baseline data at 1 year
  patients will be evaluated at 4 weeks, 8 weeks, 12 weeks, 24 weeks and 1 year after injection
Barthel Index | Change from Baseline data at 1 year
  patients will be evaluated at 4 weeks, 8 weeks, 12 weeks, 24 weeks and 1 year after injection
6 minute walking test | Change from Baseline data at 1 year
  patients will be evaluated at 4 weeks, 8 weeks, 12 weeks, 24 weeks and 1 year after injection

CONTACTS AND LOCATIONS:
Overall Officials: Pong Ya-Ping, MD, Study Chair — Rehabilitation
Locations (1):
- Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

REFERENCES:
- [Background] Yelnik AP, Bonan IV. [Post stroke hemiplegia: lower limb benefit from botulinum toxin (review)]. Ann Readapt Med Phys. 2003 Jul;46(6):281-5. doi: 10.1016/s0168-6054(03)00111-9. French. PMID 12928130
- [Background] Rivera-Dominguez M, DiBenedetto M, Frisbie JH, Rossier AB. Pes cavus and claw toes deformity in patients with spinal cord injury and multiple sclerosis. Paraplegia. 1979 Feb;16(4):375-82. doi: 10.1038/sc.1978.71. PMID 431969
- [Background] Mizel MS, Yodlowski ML. Disorders of the Lesser Metatarsophalangeal Joints. J Am Acad Orthop Surg. 1995 May;3(3):166-173. doi: 10.5435/00124635-199505000-00006. PMID 10790665
- [Background] Feeney MS, Williams RL, Stephens MM. Selective lengthening of the proximal flexor tendon in the management of acquired claw toes. J Bone Joint Surg Br. 2001 Apr;83(3):335-8. doi: 10.1302/0301-620x.83b3.11506. PMID 11341415
- [Background] Boulton AJ. Pressure and the diabetic foot: clinical science and offloading techniques. Am J Surg. 2004 May;187(5A):17S-24S. doi: 10.1016/S0002-9610(03)00297-6. PMID 15147987
- [Background] Myerson MS, Shereff MJ. The pathological anatomy of claw and hammer toes. J Bone Joint Surg Am. 1989 Jan;71(1):45-9. PMID 2913002
- [Background] Truckenbrodt H, Hafner R, von Altenbockum C. Functional joint analysis of the foot in juvenile chronic arthritis. Clin Exp Rheumatol. 1994 Sep-Oct;12 Suppl 10:S91-6. PMID 7955636
- [Background] Cyphers SM, Feiwell E. Review of the Girdlestone-Taylor procedure for clawtoes in myelodysplasia. Foot Ankle. 1988 Apr;8(5):229-33. doi: 10.1177/107110078800800501. PMID 3366427
- [Background] Bernbach EH, Bernbach MR. A box joint arthrodesis for the proximal interphalangeal joint in claw toe deformity. J Am Podiatr Med Assoc. 1985 Nov;75(11):575-80. doi: 10.7547/87507315-75-11-575. No abstract available. PMID 4067859
- [Background] Gracies JM, Elovic E, McGuire J, Simpson DM. Traditional pharmacological treatments for spasticity. Part I: Local treatments. Muscle Nerve Suppl. 1997;6:S61-91. PMID 9826983
- [Background] Gajiwala KJ, Sams SB, Pandya N, Wagh A. A new dynamic lumbrical simulating splint for claw hand deformity. Plast Reconstr Surg. 1991 Jan;87(1):170-3. doi: 10.1097/00006534-199101000-00030. PMID 1984264
- [Background] Gracies JM, Nance P, Elovic E, McGuire J, Simpson DM. Traditional pharmacological treatments for spasticity. Part II: General and regional treatments. Muscle Nerve Suppl. 1997;6:S92-120. PMID 9826984
- [Background] O'Brien CF. Treatment of spasticity with botulinum toxin. Clin J Pain. 2002 Nov-Dec;18(6 Suppl):S182-90. doi: 10.1097/00002508-200211001-00011. PMID 12569967
- [Background] Jankovic J. Botulinum toxin in clinical practice. J Neurol Neurosurg Psychiatry. 2004 Jul;75(7):951-7. doi: 10.1136/jnnp.2003.034702. PMID 15201348
- [Background] Korelitz BI, Sommers SC. Responses to drug therapy in ulcerative colitis. Evaluation by rectal biopsy and histopathological changes. Am J Gastroenterol. 1975 Nov;64(5):365-70. PMID 2008
- [Background] Stoquart GG, Detrembleur C, Palumbo S, Deltombe T, Lejeune TM. Effect of botulinum toxin injection in the rectus femoris on stiff-knee gait in people with stroke: a prospective observational study. Arch Phys Med Rehabil. 2008 Jan;89(1):56-61. doi: 10.1016/j.apmr.2007.08.131. PMID 18164331
- [Background] Lim EC, Ong BK, Seet RC. Botulinum toxin-A injections for spastic toe clawing. Parkinsonism Relat Disord. 2006 Jan;12(1):43-7. doi: 10.1016/j.parkreldis.2005.06.008. Epub 2005 Sep 29. PMID 16198612
- [Background] Suputtitada A. Local botulinum toxin type A injections in the treatment of spastic toes. Am J Phys Med Rehabil. 2002 Oct;81(10):770-5. doi: 10.1097/00002060-200210000-00009. PMID 12362118
- [Background] Chin TY, Nattrass GR, Selber P, Graham HK. Accuracy of intramuscular injection of botulinum toxin A in juvenile cerebral palsy: a comparison between manual needle placement and placement guided by electrical stimulation. J Pediatr Orthop. 2005 May-Jun;25(3):286-91. doi: 10.1097/01.bpo.0000150819.72608.86. PMID 15832139
- [Background] Molloy FM, Shill HA, Kaelin-Lang A, Karp BI. Accuracy of muscle localization without EMG: implications for treatment of limb dystonia. Neurology. 2002 Mar 12;58(5):805-7. doi: 10.1212/wnl.58.5.805. PMID 11889247
- [Background] O'Brien CF. Injection techniques for botulinum toxin using electromyography and electrical stimulation. Muscle Nerve Suppl. 1997;6:S176-80. PMID 9826989
- [Background] Berweck S, Schroeder AS, Fietzek UM, Heinen F. Sonography-guided injection of botulinum toxin in children with cerebral palsy. Lancet. 2004 Jan 17;363(9404):249-50. doi: 10.1016/S0140-6736(03)15351-2. No abstract available. PMID 14738817
- [Background] Schroeder AS, Berweck S, Lee SH, Heinen F. Botulinum toxin treatment of children with cerebral palsy - a short review of different injection techniques. Neurotox Res. 2006 Apr;9(2-3):189-96. doi: 10.1007/BF03033938. PMID 16785117
- [Background] Sconfienza LM, Perrone N, Lacelli F, Lentino C, Serafini G. Ultrasound-guided injection of botulinum toxin A in the treatment of iliopsoas spasticity. J Ultrasound. 2008 Sep;11(3):113-7. doi: 10.1016/j.jus.2008.05.002. Epub 2008 Jul 3. PMID 23396653
- [Background] Rivest J, Lees AJ, Marsden CD. Writer's cramp: treatment with botulinum toxin injections. Mov Disord. 1991;6(1):55-9. doi: 10.1002/mds.870060110. PMID 2005922
- [Background] Critchfield J. Considering the immune response to botulinum toxin. Clin J Pain. 2002 Nov-Dec;18(6 Suppl):S133-41. doi: 10.1097/00002508-200211001-00004. PMID 12569960